CLINICAL TRIAL: NCT00006025
Title: Phase I-II Trial of CPT-11 and Temozolomide (Temodar) in Patients With Recurrent Malignant Glioma
Brief Title: Temozolomide Plus Irinotecan in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: NABTC-9907; CDR0000068037 (Registry Identifier: PDQ (Physician Data Query)); UCLA-0006095; NCI-2012-02353 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of temozolomide plus irinotecan in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of irinotecan when administered with temozolomide in patients with recurrent malignant glioma.
* Determine the safety profile of this regimen in this patient population.
* Determine the efficacy of this treatment regimen as measured by 6-month progression-free survival and objective tumor response in these patients.
* Characterize the pharmacokinetics of this treatment regimen in these patients.
* Determine the antitumor activity of this treatment regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of irinotecan. Patients are stratified according to concurrent enzyme-inducing anti-epileptic drugs (EIAEDs) (e.g., phenytoin, phenobarbital, carbamazepine, or primidone) (yes vs no).

In phase I of the study, patients receive oral temozolomide on days 1-5 and irinotecan IV over 90 minutes on days 1 and 14. Treatment continues every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients concurrently on EIAEDs undergo dose escalation of irinotecan. Cohorts of 3 to 6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity.

In phase II of the study, patients receive the same treatment as in phase I at the MTD.

Patients are followed every 2 months for 1 year, every 3 months for 1 year, every 4 months for 1 year, every 6 months until progression, and then every 4 months for survival.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for phase I within 10 months and 48 patients will be accrued for phase II within 6-8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial malignant primary glioma of one of the following subtypes:

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Mixed malignant glioma
* Original histology of low-grade glioma allowed if subsequent histological confirmation of malignant glioma
* Measurable recurrent or residual primary disease by MRI

  * Lesions with clearly defined margins
* Evidence of tumor recurrence or progression by MRI or CT scan
* Confirmation of true progressive disease by PET or thallium scan, magnetic resonance spectroscopy, or surgical documentation after prior interstitial brachytherapy or stereotactic radiosurgery
* No more than 3 relapses after prior chemotherapy/cytotoxic therapy (including polifeprosan 20 with carmustine implant) for phase I and no more than 2 relapses for phase II

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No uncontrolled hypertension, unstable angina, or symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No serious uncontrolled cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No mental incapacitation
* HIV negative
* No AIDS-related disease
* No significant ongoing alcoholism or substance abuse
* No severe nonmalignant systemic disease
* No active infection
* No other severe disease that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior interferon or thalidomide and recovered
* No concurrent anticancer immunotherapy
* No concurrent sargramostim (GM-CSF)
* No concurrent prophylactic filgrastim (G-CSF) during first course of study therapy

Chemotherapy:

* See Disease Characteristics
* Recovered from prior chemotherapy
* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosourea)
* Prior radiosensitizers allowed
* No prior temozolomide or irinotecan
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* At least 1 week since prior tamoxifen and recovered
* No concurrent anticancer hormonal therapy
* Phase II:

  * Non-increasing dose of corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent anticancer radiotherapy

Surgery:

* See Disease Characteristics
* At least 1-3 weeks since prior surgical resection and recovered

Other:

* At least 1 week since prior noncytotoxic agents (e.g., isotretinoin) and recovered
* Concurrent enzyme-inducing anti-epileptic drugs with or without steroids allowed
* No concurrent valproic acid as a single agent
* No concurrent medication that would preclude study (e.g., nonsteroidal immunosuppressive agents)
* No other concurrent investigational drugs
* No concurrent participation in other clinical study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01-05 (Actual); Primary Completion 2005-01-10 (Actual); Study Completion 2007-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Kwan A. Yung, MD, Study Chair — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Loghin ME, Prados MD, Wen P, Junck L, Lieberman F, Fine H, Fink KL, Metha M, Kuhn J, Lamborn K, Chang SM, Cloughesy T, DeAngelis LM, Robins IH, Aldape KD, Yung WK. Phase I study of temozolomide and irinotecan for recurrent malignant gliomas in patients receiving enzyme-inducing antiepileptic drugs: a north american brain tumor consortium study. Clin Cancer Res. 2007 Dec 1;13(23):7133-8. doi: 10.1158/1078-0432.CCR-07-0874. PMID 18056194